CLINICAL TRIAL: NCT01675791
Title: A Dose-response Evaluation of ALK Tree AIT
Brief Title: A Dose-response Evaluation of ALK (the Sponsor) Tree Allergy Immunotherapy Tablet
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TT-02
Record Dates: First submitted 2012-08-27; First posted 2012-08-30 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Birch Pollen Allergy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- ALK tree AIT Placebo (Placebo Comparator): 1 AIT administered sublingually every day
  Interventions: Biological: ALK tree AIT Placebo
- ALK tree AIT 0.5 DU (Experimental): 1 AIT administered sublingually every day
  Interventions: Biological: ALK tree AIT 0.5 DU
- ALK tree AIT 1 DU (Experimental): 1 AIT administered sublingually every day
  Interventions: Biological: ALK tree AIT 1 DU
- ALK tree AIT 2 DU (Experimental): 1 AIT administered sublingually every day
  Interventions: Biological: ALK tree AIT 2 DU
- ALK tree AIT 4 DU (Experimental): 1 AIT administered sublingually every day
  Interventions: Biological: ALK tree AIT 4 DU
- ALK tree AIT 7 DU (Experimental): 1 AIT administered sublingually every day
  Interventions: Biological: ALK tree AIT 7 DU
- ALK tree AIT 12 DU (Experimental): 1 AIT administered sublingually every day
  Interventions: Biological: ALK tree AIT 12 DU

INTERVENTIONS:
Biological: ALK tree AIT 0.5 DU
  Arms: ALK tree AIT 0.5 DU
Biological: ALK tree AIT 1 DU
  Arms: ALK tree AIT 1 DU
Biological: ALK tree AIT 2 DU
  Arms: ALK tree AIT 2 DU
Biological: ALK tree AIT 4 DU
  Arms: ALK tree AIT 4 DU
Biological: ALK tree AIT 7 DU
  Arms: ALK tree AIT 7 DU
Biological: ALK tree AIT 12 DU
  Arms: ALK tree AIT 12 DU
Biological: ALK tree AIT Placebo
  Arms: ALK tree AIT Placebo

SUMMARY:
The primary aim of this trial is to evaluate the dose-response relationship for the ALK tree AIT administered once daily in order to define a dose-range that would be suitable for at-home administration.

ELIGIBILITY:
Inclusion Criteria:

* A history of moderate to severe birch pollen allergy
* Use of symptomatic medication for treatment of birch pollen allergy
* Positive skin prick test to birch extract
* Positive specific IgE against Bet v 1

Exclusion Criteria:

* Overlapping perennial allergies
* History of uncontrolled asthma within the last 3 months
* FEV1 < 70% of predicted value in adults or FEV1 < 80% of predicted value in adolescents
* Previous or ongoing treatment with immunotherapy

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 637 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Allergy symptom severity scores on a scale from 0-3 | During the birch pollen season 2013, an expected average of 3 weeks
  Determine the dose-efficacy response relationship of the ALK tree AIT. This information will, in combination with the evaluation of the frequency and severity of adverse events, form the basis of the conclusion on the primary endpoint.
Adverse events frequency | Throughout the trial, an expected average of 8 months
  Determine the dose-safety response relationship of the ALK tree AIT. This information will, in combination with the evaluation of the allergy symptoms, form the basis of the conclusion on the primary endpoint.

SECONDARY OUTCOMES:
Adverse events severity | Throughout the trial, an expected average of 8 months
  Determine the dose-safety response relationship of the ALK tree AIT. This information will, in combination with the evaluation of the allergy symptoms, form the basis of the conclusion on the primary endpoint.

CONTACTS AND LOCATIONS:
Locations (2):
- Skin and Allergy Hospital, Helsinki University Central Hospital, Helsinki, HUS, Finland
- Slotervaart Ziekenhuis, Amsterdam, Netherlands